CLINICAL TRIAL: NCT00547417
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Tadalafil Administered "On Demand" to Men of Various Populations With Erectile Dysfunction
Brief Title: To Determine Effect and Safety of Tadalafil Taken by Men of Different Races and With Different Diseases When Needed for Erections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7006; H6D-MC-LVFN
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): tadalafil
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 20 mg tadalafil tablet taken by mouth, as needed, no more than once a day, for 12 weeks.
  Other Names: LY450190; Cialis; IC351

SUMMARY:
To compare men of different races and those with diabetes or depression to white men that do not have diabetes or depression but also suffer from the inability to get or keep an erection.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months history of erectile dysfunction (ED)
* Anticipate a monogamous relationship with a female sexual partner
* Be able to make minimum required sexual intercourse attempts
* Abstain from using any other ED treatment

Exclusion Criteria:

* Other primary sexual disorders
* History of penile implant or clinically significant penile deformity
* History or current nitrate use
* History of certain heart problems
* History of certain kidney problems

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1933 (Actual)
Dates: Start 2003-07; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Change in the scores of the IIEF scale's Erectile Function domain, questions 1-5 and 15 | 12 weeks

SECONDARY OUTCOMES:
Percentage of Yes answers to questions 2 and 3 of the Sexual Encounter Profile | 12 weeks
Evaluation of score changes for selected GAQ, PAIRS, and IIEF questions. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com